CLINICAL TRIAL: NCT02138513
Title: (Cost-) Effectiveness of Mindfulness Based Cognitive Therapy (MBCT) in Cancer Patients: a Superiority Trial of Online and Face-to-face Treatment Versus Treatment as Usual (TAU).
Brief Title: (Cost-)Effectiveness of Mindfulness-Based Cognitive Therapy (MBCT) in Cancer Patients
Acronym: BeMind
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2012.WO14.C153; NL46338.091.13 (Registry Identifier: Toetsingonline)
Record Dates: First submitted 2014-05-06; First posted 2014-05-14 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2016-02

CONDITIONS: Distress; Anxiety; Depression
Keywords: Mindfulness; MBCT; Cancer; Oncology; E-health; Cost-effectiveness
MeSH Terms: conditions — Anxiety Disorders; Depression; Neoplasms | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Online MBCT (Experimental)
  Interventions: Behavioral: Mindfulness Based Cognitive Therapy
- group MBCT (Experimental)
  Interventions: Behavioral: Mindfulness Based Cognitive Therapy
- Treatment as usual (No Intervention): 3 months waiting list, subsequent assignment to group or online MBCT

INTERVENTIONS:
Behavioral: Mindfulness Based Cognitive Therapy — This MBCT protocol consists of 8 weekly sessions of 2,5 hours each and a silent day of 6 hours of meditation practice. Similar to group MBCT, in the online MBCT group, participants will be asked to practice at home for 45 minutes, 6 days a week. They will receive files with meditation and yoga exercises to support this.
  Arms: Online MBCT; group MBCT

SUMMARY:
Mindfulness-based cognitive therapy has been demonstrated to be effective in reducing anxiety, depression and fatigue in cancer patients. As this intervention can be offered in groups, costs are relatively low. In addition, delivering MBCT online might make the intervention more accessible and cost-effectiveness. However, more information is needed about what treatment works best for which patient.

Therefore, the aim of this study is to investigate clinical and cost-effectiveness of both individual MBCT online and MBCT offered as a group training compared to TAU .

Study design: The design of the study will be a multi-centre, randomised, superiority trial, comparing MBCT online and MBCT offered as a group training with TAU. Participants in the TAU condition will be randomised to one of the treatment conditions after 3 months. Main assessments will take place at baseline (T0), post-treatment (T1), and 3 (T2) and 9 months after post-treatment (T3).

We expect the MBCT conditions to be superior to TAU in terms of improving mindfulness skills, anxiety and depressive compants, psychological well-being, rumination and fear of cancer recurrence. We also expect the MBCT to result in patients returning to work earlier, have a higher work ability and have lower medical care costs, thereby being more cost-effective than TAU.

ELIGIBILITY:
Inclusion Criteria:

* HADS ≥ 11
* Cancer diagnosis (at present or past)
* Stable dose if using psychopharmacological medication for at least 3 months
* computer literacy and acces to internet
* capable of filling out questionnaires in Dutch

Exclusion Criteria:

* severe psychiatric morbidity as psychoses, suicidal ideation
* previous mindfulness-based treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2014-04; Primary Completion 2016-07-20 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in anxiety and depressive symptoms | 0 (baseline), 3 months (post intervention)
  Anxiety and depressive symptoms as assessed by the Hospital Anxiety and Depression-scale (HADS). The HADS is a self-report questionnaire that comprises 14 items measuring feelings of generalized fear and depressive symptoms. The HADS is considered a reliable and valid instrument for assessing anxiety and depression in medical patients and is sensitive to change (Herrmann, 1997; Bjelland et al., 2002). This instrument was also validated in a palliative cancer population (Akechi, 2006).

SECONDARY OUTCOMES:
Change from baseline in fear of cancer recurrence | 0, 3 (post intervention), 6 (3mo follow-up) and 12 months (9mo follow-up)
  Fear of cancer recurrence will be assessed with the Fear of Cancer Recurrence Inventory (FCRI; Simard & Savard, 2009a; van der Lee et al., 2012).
DSM-IV Axis I mood or anxiety disorders | 0, 3 (post intervention), 12 months (9mo follow-up)
  DSM IV Axis I psychiatric disorder as diagnosed by a structured interview
Change from baseline in positive mental health | 0, 3 (post intervention), 6 (3mo follow-up) and 12 months (9mo follow-up)
  The Mental Health Continuum-Short Form (MHC-SF) measures positive mental health and comprises 14 items, representing various feelings of well-being. Respondents rate the frequency of every feeling in the past month on a 6-point Likert scale (never, once or twice a month, about once a week, two or three times a week, almost every day, every day). The MHC-SF contains three subscales: emotional, psychological and social well-being. MHC-SF has shown high internal and moderate test-retest reliability, convergent and discriminant validity.
Change from baseline in healthcare consumption | 0, 3 (post intervention), 6 (3mo follow-up) and 12 months (9mo follow-up)
  The TIC-P generates quantitative data about direct medical costs and indirect societal costs as a consequence of psychological/psychiatric illnesses.
Change from baseline in health-related quality of life | 0, 3 (post intervention), 6 (3mo follow-up) and 12 months (9mo follow-up)
  To measure the quality of the health status of cancer patients a validated health-related quality of life (HRQoL) instrument will be used, the EuroQol-5D (EQ-5D). This HRQoL instrument will be completed by the patient together with a researcher and is available in a validated Dutch translation (Lamers, 2005). The EQ-5D is a generic HRQoL instrument comprising five domains: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The EQ-5D index is obtained by applying predetermined weights to the five domains. This index gives a societal-based global quantification of the participant's health status on a scale ranging from 0 (death) to 1 (perfect health). Participants will also be asked to rate their overall HRQoL on a visual analogue scale (EQ- 5D VAS) consisting of a vertical line ranging from 0 (worst imaginable health status) to 100 (best imaginable).
Change from baseline in health-related quality of life | 0, 3 (post intervention), 6 (3mo follow-up) and 12 months (9mo follow-up)
  In addition to the EQ-5D, the SF-12 will be administered for explorative purposes for there are indications that the SF-12 is more sensitive for changes in HRQol in populations with less severe morbidity (Johnson and Coons, 1998).
Change from baseline in mindfulness skills | 0, 3 (post intervention), 6 (3mo follow-up) and 12 months (9mo follow-up)
  The 39-item Five Facet Mindfulness Questionnaire has been developed as a reliable and valid comprehensive instrument for assessing different aspects of mindfulness. A Dutch 24-item short form of the FFMQ (FFMQ-SF) was developed and assessed in a sample of 376 adults with clinically relevant symptoms of depression and anxiety and cross-validated in an independent sample of patients with fibromyalgia. Confirmatory factor analyses showed good model fit for the five-factor structure of the FFMQ-SF: observing, describing, acting with awareness, nonjudging, and nonreactivity. The FFMQ-SF was related to measures of psychological symptoms, well-being, experiential avoidance, and the personality factors neuroticism and openness to experience.
Change from baseline in rumination | 0, 3 (post intervention), 6 (3mo follow-up) and 12 months (9mo follow-up)
  The rumination subscale of the RRQ assesses a neurotic self-attentiveness (i.e. recurrent, primarily past-oriented thinking about the self), which is prompted by threats, losses, of injustices to the self. Subjects rate their level of agreement of disagreement on a five-point rating scale (e.g., "I always seem to be rehashing in my mind recent things I've said or done"). There is evidence of good internal consistency (.90) and stability over a 10-month period and convergent validity. The measure in the current study was translated into Dutch using the guidelines of the International Test Commission (Hambleton, 1994). Cronbach's alphas were .88 and .90 in Sample 1, and .90 and .91 in Sample 2, respectively (Luyckx et al., 2008).
Change from baseline in personality assessment | 0 (baseline) and 12 months (9mo follow-up)
  Personality is measured with the NEO Five Factor Inventory (NEO-FFI, Costa & McCrae, 1992) which consists of five domains: neuroticism, extraversion, openness, altruism, and conscientiousness.
Change in mindfulness skills during intervention | week 2,3,4,5,6,7,8 and 9 of intervention
  The Mindful Attention Awareness Scale (MAAS) will be administered before each MBCT session to assess mindful attention in daily life
Group cohesion during intervention | week 4 and week 9 during intervention
  We will examine self-reported individual group cohesion ratings during the MBCT training with a Dutch Group Cohesion Questionnaire that has been used in cancer patients before (May et al., 2008). The GCQ-23 uses 22 items across four scales: the bond with the group as whole, the bond with other members, cooperation within the group and the instrumental value. Each item is rated from 1 (totally disagree) to 6 (totally agree). Internal consistency of all scales was reported to range from adequate to good (0.66-0.88).
Working alliance during intervention | week 4 and week 9 during intervention
  The Working Alliance Inventory (WAI) is most often used to assess working alliance between participant and healthcare professional. We will use the Dutch translation of the short form (WAI-S, Vervaeke & Vertommen, 1996), which is closely related to the original scale and also has good psychometric and predictive quality (Busseri & Tyler, 2003). The WAI-S is a 12 item, self report questionnaire, rated on a 7-point Likert scale (1 = never to 7 = always) with three subscales: 1) agreement between participant and therapist on the goals of the therapy; 2) agreement on the rationale of the therapy addressing the problems of the participant; and 3) the quality of the interpersonal bond between the participant and the therapist.
Change in mood during intervention | week 2,3,4,5,6,7,8 and 9 of intervention
  In the current study, positive and negative affect is assessed before each MBCT session using the International Positive and Negative Affect Scale - Short Form. The cross-sample stability, internal reliability, temporal stability, crosscultural factorial invariance, and convergent and criterion-related validities of the I-PANAS-SF were examined and found to be psychometrically acceptable (Thompson, 2007).
Change from baseline in anxiety and depressive symptoms - follow up | 0, (baseline) 6 (3mo follow-up) and 12 months (9mo follow-up)
  Hospital Anxiety and Depression Scale - anxiety and depressive symptoms at follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Anne EM Speckens, MD, PhD, Principal Investigator — Radboud University Medical Centre Nijmegen
Locations (2):
- Netherlands (2):
  - Radboud University Medical Centre for Mindfulness, Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland
  - Helen Dowling Institute, Bilthoven, Utrecht

REFERENCES:
- [Derived] Bisseling EM, Compen FR, Schellekens MPJ, Thewes B, Speckens AEM, van der Lee ML. Exploring Fear of Cancer Recurrence in a Sample of Heterogeneous Distressed Cancer Patients with and Without a Psychiatric Disorder. J Clin Psychol Med Settings. 2021 Sep;28(3):419-426. doi: 10.1007/s10880-021-09776-2. Epub 2021 Jun 17. PMID 34138447
- [Derived] Bisseling E, Cillessen L, Spinhoven P, Schellekens M, Compen F, van der Lee M, Speckens A. Development of the Therapeutic Alliance and its Association With Internet-Based Mindfulness-Based Cognitive Therapy for Distressed Cancer Patients: Secondary Analysis of a Multicenter Randomized Controlled Trial. J Med Internet Res. 2019 Oct 18;21(10):e14065. doi: 10.2196/14065. PMID 31628791
- [Derived] Compen F, Bisseling E, Schellekens M, Donders R, Carlson L, van der Lee M, Speckens A. Face-to-Face and Internet-Based Mindfulness-Based Cognitive Therapy Compared With Treatment as Usual in Reducing Psychological Distress in Patients With Cancer: A Multicenter Randomized Controlled Trial. J Clin Oncol. 2018 Aug 10;36(23):2413-2421. doi: 10.1200/JCO.2017.76.5669. Epub 2018 Jun 28. PMID 29953304
- [Derived] Compen FR, Bisseling EM, Van der Lee ML, Adang EM, Donders AR, Speckens AE. Study protocol of a multicenter randomized controlled trial comparing the effectiveness of group and individual internet-based Mindfulness-Based Cognitive Therapy with treatment as usual in reducing psychological distress in cancer patients: the BeMind study. BMC Psychol. 2015 Aug 13;3(1):27. doi: 10.1186/s40359-015-0084-1. eCollection 2015. PMID 26273472